CLINICAL TRIAL: NCT03922477
Title: A Phase Ib, Open-Label Study Evaluating the Safety and Pharmacokinetics of Atezolizumab (Anti-PD-L1 Antibody) Administered in Combination With Hu5F9-G4 to Patients With Relapsed and/or Refractory Acute Myeloid Leukemia
Brief Title: A Study Evaluating the Safety and Pharmacokinetics of Atezolizumab Administered in Combination With Hu5F9-G4 to Patients With Relapsed and/or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor decided to discontinue the development of atezolizumab in combination with magrolimab in the AML indication.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO40828
Record Dates: First submitted 2019-04-11; First posted 2019-04-22 (Actual); Results first posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — atezolizumab; magrolimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + Hu5F9-G4 (Experimental): An initial safety evaluation will be performed in participants with relapsed AML. If atezolizumab in combination with Hu5F9-G4 is initially safe and tolerable in participants an additional cohort with R/R AML will be evaluated to further test the safety and anti-tumor activity. If dose-limiting toxicities (DLT) are observed in >=33% of participants in this initial cohort, a dose de-escalation cohort will be enrolled. If less than 33% of enrolled and dosed participants in any given cohort experience a DLT, an expansion cohort of 15 participants will be enrolled at the highest tolerated dose for this combination. If a dose de-escalation cohort is needed, an expansion cohort will be enrolled at the lower tolerated dose for this combination.
  Interventions: Drug: Atezolizumab; Drug: Hu5F9-G4

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered to participants by IV infusion at a fixed dose starting on Day 22 of Cycle 1. In subsequent cycles (Cycles 2 and beyond), IV atezolizumab will be given every 2 weeks (Q2W) on Days 8 and 22 of each 28-day cycle.
  Other Names: Tecentriq
Drug: Hu5F9-G4 — Two priming doses of 1 mg/kg of Hu5F9-G4 will be administered to participants by continuous IV infusion on Days 1 and 4 of Cycle 1, followed by loading doses of 15 mg/kg IV on Day 8 and 30 mg/kg IV on Day 11. Starting on Day 15 of Cycle 1, Hu5F9-G4 maintenance will be given by IV infusion at a dose of 30 mg/kg once a week (QW) of each 28-day cycle. Dosing for de-escalation, if needed: Hu5F9-G4 will be given as two priming doses of 1 mg/kg IV on Days 1 and 4, followed by loading doses of 10 mg/kg IV on Day 8 and 15 mg/kg on Day 11. Starting on Day 15, maintenance treatment with Hu5F9-G4 will be given by IV infusion at a dose of 15 mg/kg once a week (QW).

SUMMARY:
This Phase Ib study is designed to evaluate the safety and pharmacokinetics of atezolizumab when given in combination with Hu5F9-G4 to patients with relapsed or refractory (R/R) acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group Performance Status 0-2
* Documented and confirmed R/R AML per WHO classification, except acute promyelocytic leukemia, and lack of response to all therapies of known benefit
* Adequate end-organ function
* Negative HIV test at screening
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by quantitative hepatitis B virus (HBV) DNA <500 IU/mL at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening
* Willingness and ability to provide pretreatment bone marrow aspirate and biopsy and agreement to provide subsequent bone marrow aspirates and biopsies during study treatment
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm
* For women who are not postmenopausal or surgically sterile: requirement for a negative serum pregnancy test result within 14 days prior to initiation of study treatment

Exclusion Criteria:

* Previous allogeneic hematopoietic stem cell transplant within 6 months prior to enrollment, active graft versus host disease, or requiring transplant-related immunosuppression
* Prior solid organ transplant
* Evidence of active central nervous system (CNS) involvement by leukemia
* Pregnancy or lactation or intention to become pregnant during the study or within 5 months after the final dose of atezolizumab and/or Hu5F9-G4, whichever is longer
* History of idiopathic pulmonary fibrosis, organizing pneumonitis, drug-induced pneumonitis, or idiopathic pneumonitis
* History of autoimmune disease. Patients with a history of autoimmune-related hypothyroidism who are on a stable dose of thyroid replacement may be eligible for this study. Patients with controlled Type 1 diabetes mellitus who are on a stable insulin regimen may be eligible for this study. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are eligible for the study provided all of the following conditions are met: (1) Rash must cover <10% of body surface area, (2) Disease is well controlled at baseline and requires only low-potency topical corticosteroids, (3) No occurrence of acute exacerbations of the underlying condition that require psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
* Treatment with investigational therapy within 14 days prior to initiation of study drug
* Any approved AML-related therapy within 14 days prior to enrollment. Granulocyte colony-stimulating factor to treat neutropenic fever and/or infection is permitted. Hydroxyurea may be used throughout the trial to control peripheral blood blast counts in response to the first dose of study treatment and during the first 4 weeks of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Yale, New Haven, Connecticut
  - Columbia University, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Atezolizumab + Hu5F9-G4: An initial safety evaluation was performed in participants with relapsed AML. If atezolizumab in combination with Hu5F9-G4 was initially safe and tolerable in participants an additional cohort with R/R AML was to be evaluated to further test the safety and anti-tumor activity. Atezolizumab was administered to participants by IV infusion at a fixed dose of 840 mg starting on Day 22 of Cycle 1. In subsequent cycles, IV atezolizumab was given every 2 weeks (Q2W) on Days 8 and 22 of each 28-day cycle. Two priming doses of 1 mg/kg of Hu5F9-G4 were administered to participants by continuous IV infusion on Days 1 and 4 of Cycle 1, followed by loading doses of 15 mg/kg IV on Day 8 and 30 mg/kg IV on Day 11. Starting on Day 15 of Cycle 1, Hu5F9-G4 maintenance was given by IV infusion at a dose of 30 mg/kg once a week (QW) of each 28-day cycle.
Period: Overall Study
Arm/Group | Atezolizumab + Hu5F9-G4
Started | 13
Completed | 0
Not Completed | 13
Not completed — Death | 9
Not completed — Fall leading to death prior to treatment initiation. | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of participants with at least one adverse event.
Time Frame: Up to approximately 13 months after first participant enrolled
Population: Safety population included all participants with any amount of either study drug, with participants grouped as a whole.
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 11
Percentage of participants | 100

2. Primary Outcome: Complete Remission (CR)
Description: The CR rate is assessed as the percentage of participants who achieve a CR, complete remission with incomplete platelet recovery (CRp), complete remission with incomplete hematologic recovery (CRi), or complete remission with partial hematologic recovery (CRh) (as defined by the IWG 2003 and ELN 2010 criteria) after up to six cycles of combination therapy.
Time Frame: Up to approximately 3 months after first participant enrolled
Population: The efficacy analysis population included all participants who received any amount of either study drug, with participants grouped as a whole.
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 11
Percentage of participants | 0

3. Primary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the initial response (CR, CRp, CRi, CRh, or partial remission [PR]) to the time of disease progression or death, whichever occurs first
Time Frame: Up to approximately 3 months after first particpant enrolled
Population: The efficacy analysis population included all participants who received any amount of either study drug, with participants grouped as a whole. No participants were analyzed because no participants responded.
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 0

4. Secondary Outcome: Serum Concentrations of Atezolizumab
Description: C=cycle (cycle=28 days) ; D=day; PTFI=prior to first infusion; TDV=treatment discontinuation visit; UTA=up to approximately; M=month
Time Frame: C1 D22 PTFI of Hu5F9-G4 and atezolizumab, and 30 minutes after atezolizumab infusion; C2 D8 PTFI; C2 D22 PTFI; C3 D22 PTFI; C4 D22 PTFI; C8 D22 PTFI; C12 D22 PTFI; C16 D22 PTFI; TDV (up to C16 D21);120 days after final dose of atezolizumab (UTA 37M)
Population: Samples for PK analysis were collected, but due to the small number of participants which reduces the scientific merit of any analysis no PK assays were performed and samples were discarded, hence no PK data are available.
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 0

5. Secondary Outcome: Serum Concentrations of Hu5F9-G4
Description: C=cycle (cycle=28 days); D=Day; PTFI=prior to first infusion; H=hour; AEOI=after end of infusion; TDV=treatment discontinuation visit; UTA=up to approximately; M=months; E=every; T=thereafter
Time Frame: C1D1 PTFI&1H AEOI; C1D8 PTFI,&1H AEOI; C1D11 PTFI,&1H AEOI; C1D22 1H AEOI; C2D1 PTFI,&1H AEOI; C2D8 PTFI; C3D1 PTFI,&1H AEOI; C5D1 PTFI; C7D1 PTFI, C9D1 PTFI; C11D1 PTFI; C13D1 PTFI; C15D1 PTFI; C17D1&D1 E 2C T PTFI(UTA 37M);TDV(up to C16D21)(UTA 37M)
Population: as for outcome 4
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 0

6. Secondary Outcome: Objective Response Rate
Description: Objective response rate is defined as the percentage of participants with a partial remission (PR) or better (i.e., CR + CRp + CRi + CRh+ PR).
Time Frame: Up to approximately 3 months after first participant enrolled
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 11
Percentage of participants | 0

7. Secondary Outcome: Event-Free Survival
Description: Event-free survival is defined as the time from study entry to the date of induction treatment failure or relapse from CR, CRp, CRh, CRi, or death from any cause.
Time Frame: Up to approximately 3 months after first participant enrolled
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 11
Months | 1.7 [1.02 to 2.83]

8. Secondary Outcome: Leukemia-Free Survival
Description: Leukemia-free survival is defined (only for participants achieving a CR, CRp, CRh, or CRi) as the time from the date of achievement of remission (CR, CRp, or CRi) until the date of relapse from CR, CRp, CRh, CRi, or death from any cause.
Time Frame: Up to approximately 3 months after first participant enrolled
Population: No participants were analyzed because no participants received an objective response.
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 0

9. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from study entry to the date of death from any cause.
Time Frame: Up to approximately 13 months after first participant enrolled
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 11
Months | 4.1 [1.74 to 6.37]

10. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (Investigator) is defined as the time from the first day of study treatment to disease progression or death, whichever occurs first.
Time Frame: Up to approximately 3 months after first participant enrolled
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 11
Months | 2.8 [1.48 to 3.02]

11. Secondary Outcome: Rate of Transfusion Independence
Description: Rate of transfusion independence is defined as the percentage of participants who achieve transfusion independence (i.e., achieving any continuous 56-day window without requiring platelet or RBC transfusions) at any time during study treatment.
Time Frame: Up to approximately 3 months after first participant enrolled
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 11
Percentage of participants | 0

12. Secondary Outcome: Duration of Transfusion Independence
Description: Duration of transfusion independence is defined as the number of consecutive days of transfusion independence, measured from 1 day after the last transfusion to disease progression or subsequent transfusion.
Time Frame: Up to approximately 3 months after first participant enrolled
Population: None of the participants achieved transfusion independence, hence duration of independence was not calculated.
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 0

13. Secondary Outcome: Incidence of Anti-Drug Antibodies (ADAs) Against Atezolizumab During the Study Relative to the Prevalence of ADAs at Baseline
Time Frame: Baseline up to approximately 37 months
Population: Samples for ADA analysis were collected, but due to the small number of participants which reduces the scientific merit of any analysis no ADA assays were performed and samples were discarded, hence no ADA data are available.
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 0

14. Secondary Outcome: Incidence of ADAs Against Hu5F9-G4 During the Study Relative to the Prevalence of ADAs at Baseline
Time Frame: Baseline up to approximately 37 months
Population: as for outcome 13
Arm/Group | Atezolizumab + Hu5F9-G4
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 3 November 2020 (approximately 13 months)
Description: Safety population included all participants with any amount of either study drug, with participants grouped as a whole.
Groups:
- Safety_Cohort: An initial safety evaluation was to be performed in participants with relapsed AML. A total of 19 participants were screened for enrollment; 8 failed screening. 13 were enrolled but only 11 received study treatment. All 11 patients enrolled in the safety cohort discontinued the study.
Arm/Group | Safety_Cohort
All-Cause Mortality (participants affected / at risk) | 9/11
Serious Adverse Events (participants affected / at risk) | 10/11
Other Adverse Events (participants affected / at risk) | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety_Cohort (N=11)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Pneumonia (Infections and infestations) | 5 (9)
Sepsis (Infections and infestations) | 1 (2)
Skin infection (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety_Cohort (N=11)
Anaemia (Blood and lymphatic system disorders) | 5 (11)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Localised oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 4 (5)
Pyrexia (General disorders) | 3 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 2 (4)
Human rhinovirus test positive (Investigations) | 1 (1)
Liver function test increased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Lethargy (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Haematoma (Vascular disorders) | 1 (3)
Hypertension (Vascular disorders) | 2 (3)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT03922477/Prot_SAP_000.pdf